CLINICAL TRIAL: NCT06273072
Title: Metformin IN Asthma for Overweight and Obese Individuals (MINA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Baylor College of Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00409080; R34HL166438-01A1 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Asthma; Asthma Chronic; Overweight and Obesity
MeSH Terms: conditions — Asthma; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin hydrochloride extended-release tablets (Active Comparator): Metformin hydrochloride extended-release tablets 2000 mg once daily
  Interventions: Drug: Metformin hydrochloride extended-release tablets
- Visually identical placebo tablets (Placebo Comparator): Placebo tablet once daily
  Interventions: Drug: Visually identical placebo Metformin hydrochloride extended-release tablets

INTERVENTIONS:
Drug: Metformin hydrochloride extended-release tablets — titrated to 2000 mg once daily
  Arms: Metformin hydrochloride extended-release tablets
Drug: Visually identical placebo Metformin hydrochloride extended-release tablets — placebo
  Arms: Visually identical placebo tablets

SUMMARY:
This is a randomized clinical trial of metformin among overweight or obese adults with not well-controlled asthma despite maintenance inhaler therapy.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, parallel-arm pilot clinical trial. Adult participants who are overweight or obese and have not well-controlled asthma despite use of an inhaled corticosteroid will be randomized to metformin, an FDA-approved medication for the treatment of type 2 diabetes mellitus, or to placebo, to be taken daily for a total duration of six months. Recruitment will occur at two sites in the United States.

Randomized participants will have regular telemedicine visits to assess side effects and adherence. Additionally, participants will have a measurement of asthma outcomes at randomization and at 3 and 6 months after randomization.

The purpose of this study is to determine feasibility to inform a future multi-center clinical trial of metformin in this population.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma on maintenance therapy
* Not well-controlled asthma (ACT score <20, or at least one asthma exacerbation requiring corticosteroids in the prior 12 months)
* Overweight or obesity: Body mass index ≥25kg/m2
* Adult: Age ≥18

Exclusion Criteria:

* Currently pregnant, expect to become pregnant in the next 6 months or are currently breastfeeding
* Major cardiovascular disease: heart failure, heart attack or stroke within the last 6 months
* Other chronic lung disease, inclusive of chronic obstructive pulmonary disease, bronchiectasis, interstitial lung disease, pulmonary fibrosis
* Active smoking or former smoker with ≥20 pack-year smoking history
* Chronic kidney disease: estimated glomerular filtration rate ≤60 mL/min/1.73 m2
* Heavy alcohol use: in a typical week, 8 or more drinks for a woman or 15 or more drinks for a man
* Liver disease: elevation in aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2x the upper limit of normal or prior diagnosis of liver disease
* Anemia: hemoglobin < 13 g/dl in males and hemoglobin < 11 g/dl in females
* Taking Glucagon Like Peptide 1(GLP-1) medications for weight loss
* Diabetes (Hemoglobin A1C ≥ 6.5% or taking metformin or other medications used to treat diabetes)
* Participation in any other clinical trial (observational studies are permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of completed telemedicine visits | Baseline to week 24
  Number of participants completing at least 3 out of the 4 monitoring telemedicine visits
Adherence to study drug | Baseline to week 24
  Adherence will be measured by pill count
Retention rate | Baseline to week 24
  Investigators will collect data on the number of subjects screened, randomized, and complete the final in-person visit

SECONDARY OUTCOMES:
Asthma control as assessed by the Asthma Control Test (ACT) score | Baseline to week 24
  Difference in Asthma Control Test (ACT) score at week 24; range is from 5-25 with higher being better asthma control
Change in Asthma exacerbations rate | Baseline to week 24
  Change in (annualized) asthma exacerbations rate at week 24
Pre-bronchodilator lung function | Baseline to week 24
  Difference in volume of air exhaled in the first second during spirometry (FEV1) at week 24
Fractional exhaled nitric oxide (FeNO) | Baseline to week 24
  Difference in FeNO between baseline and week 24
Airways hyperresponsiveness | Baseline to week 24
  Difference in cumulative dose of mannitol required to precipitate a significant decrement in FEV1 between baseline at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Meredith C McCormack, M.D., M.H.S., Principal Investigator — Johns Hopkins University; Tianshi D Wu, M.D., M.H.S., Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Baylor College of Medicine, Houston, Texas